CLINICAL TRIAL: NCT03545698
Title: Enhancing and Scaling a High-Touch Home-based Primary Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Gary and Mary West Health Institute (Other)
Responsible Party: Principal Investigator, Karen Abrashkin, Medical Director, House Calls, Northwell Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-0244-NH
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Satisfaction, Consumer; Caregiver Stress
MeSH Terms: conditions — Consumer Behavior; Caregiver Burden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention (Active Comparator)
  Interventions: Other: Avizia Telehealth Platform
- Non-Telehealth Intervention (No Intervention)

INTERVENTIONS:
Other: Avizia Telehealth Platform — Avizia will be utilized as a communication tool between home-based caregivers (family members, formal caregivers, or informal caregivers) and the House Calls care management team.
  Arms: Telehealth Intervention

SUMMARY:
The overall goal of the West Health Institute-Northwell PRP is to identify a clinical and economic model that can support scaling the Northwell House Calls program within a four year implementation period, while maintaining the same level of quality, patient/caregiver satisfaction, and "high touch" provider-patient communication that the program is known for. The Clinical Trial portion of this study refers to the secondary endpoint listed below.

DETAILED DESCRIPTION:
Primary Endpoint: Northwell's House Calls program will be effectively scaled to maintain a patient census of 2000 without compromising patient and caregiver satisfaction.

Secondary Endpoint: The telehealth platform, Avizia, effectively improves communication of patient and caregiver needs to House Calls staff, and overall program satisfaction.

In order to achieve the secondary endpoint, a telehealth platform will be implemented that will allow patients and their caregivers to teleconference with their care manager, who is either a nurse or a social worker, replacing a typical visit which is completed telephonically.

Hypotheses to be tested through a home based telehealth intervention :

* Maintain longitudinal non-inferiority of: in-person acute care home visits from a provider, in-person acute care home visits from a care manager, hospitalizations, ED visits, Community Paramedicine deployments, Community Paramedicine transports to hospital, the patient's acuity level, LACE Score, Charelson Co-Morbidity score and the total number of ADLs group compared to usual care group.
* Telehealth acceptability
* decrease caregiver stress
* Improve program satisfaction
* Improve staff satisfaction and engagement

ELIGIBILITY:
Inclusion Criteria:

* Patients from the chronic and complex phone-only acuity level, from House Calls, Advanced Illness Management, Northwell Health Solutions.
* If possible, we will recruit both patient and caregiver dyads.
* The caregiver can be a family member or a paid caregiver.
* If patients are cognitively impaired, then they must have a caregiver who can verbally confirm that they will be present with the patient for the telehealth visit. -Caregiver must be present during Avizia enrollment with the research staff to ensure proper use of the device.
* The eligible patient or the eligible caregiver, must have a mobile phone number or email address listed in Allscripts is the associated chart, in order to participate in an Avizia visit with House Calls.
* Patients will be able to participate in the study regardless of cognitive impairment, if they have a caregiver who is able to consent on their behalf. This caregiver must be their power of attorney or family member, but does not have the be the caregiver present for the Avizia visit.

Exclusion Criteria:

* Patients under 18
* Patients that are cognitively impaired and unable to use the device, who also do not have a present and willing caregiver who can use the device.
* If the patient and willing caregiver do not have an email address or phone number listed on the associated chart on Allscripts.
* Patient or caregiver does not have a smart phone, tablet, laptop or desktop computer able to launch Avizia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Telehealth Acceptability Among Geriatric, Homebound patients | 12 months
  The proportion of geriatric patients who agree to use telehealth for a care management visit in lieu of a phone call visit, out of those who are offered the service.

SECONDARY OUTCOMES:
Telehealth Completion Success | 12 months
  The proportion of telehealth visits that are completed successfully, out of those that are scheduled.
Telehealth Satisfaction Among Geriatric Patients | 12 months
  The sum and average of scores across domains on the Telemedicine Satisfaction Questionnaire.
Telehealth Satisfaction Among RNs and Social Workers | 12 months
  The sum and average of scores across domains on the Telemedicine Satisfaction Questionnaire, adapted from original use with providers to use with care management staff (RNS and Social Workers).

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Smith, MD MPP, Principal Investigator — Northwell Health Solutions
Locations (1):
- Northwell Health Solutions, Advanced Illness Management, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No